CLINICAL TRIAL: NCT00457093
Title: A Double Blind, Randomized, Parallel, Cross-Over Comparision of Glycemic Control Achieved With Once a Day Insulin Glargine Versus Detemir in Type 2 Diabetes
Brief Title: A Comparison Between Glargine and Detemir Insulin in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diabetes Care Center (Industry)
Collaborators: Novo Nordisk A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06-07
Record Dates: First submitted 2007-04-03; First posted 2007-04-05 (Estimated); Last update posted 2010-11-18 (Estimated); Status verified 2007-04

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; continuous glucose monitoring; basal insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: glargine
Drug: detemir

SUMMARY:
The purpose of this study that when studies using our method of dosing adjustments driven by continuous glucose monitoring and because of the less variable glycemic effect of insulin detemir, insulin detemir treated subjects will spend a significantly greater time in the glucose target range than insulin glargine.

DETAILED DESCRIPTION:
Todate, most studies have compared insulin detemir and glargine to NPH and not to each other. Depending of their design, these studies have shown both insulins lower the fasting glucose, A1c, the incidence of hypoglycemia and are associated with less weight gain than NPH. In the only direct comparison study of these two basal insulins, insulin detemir demonstrated significantly less day to day variation than glargine as measured by glucose infusion rated during an euglycemic clamp study. Given the same incidence of hypoglycemia, this last study would suggest that insulin detemir treatment could achieve target glucose control more than glargine. We have used continuous glucose monitoring (CGMS) extensively in our practice. CGMS is arguably the most sensitive method for detecting differences in glycemic control in the outpatient setting and there by allowing fine adjustments in insulin treatment. When comparing insulin glargine to preprogrammable basal insulin as delivered by continuous subcutaneous infusion and using CGMS, we have shown significantly better glucose control with continuous subcutaneous infusion, We have also developed a method of daily insulin dosage adjustments during a continuous CGMS study from daily glucose tracings downloaded. This allows for an even more accurate basal insulin replacement per set glycemic goal. This protocol addresses a comparison of insulin glargine and insulin detemir for patients evaluated by CGMS.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* Currently on a basal insulin, that is, NPH, glargine or detemir
* Capable of self monitoring glucose >4/day
* Previously complaint with clinical recommendations
* Subject may be on oral antiglycemic medications but no change in treatment is permitted during study.

Exclusion Criteria:

* Hb A1c >9.0%
* Urinary ketosis
* Currently or expected alteration in insulin sensitivity such as major surgery, infection, renal failure (creatine >1.5 mg/dL) glucocorticoid treatment, recent (within 2 weeks) serious hypoglycaemic episode (requires assistance of another)
* Currently participating in another clinical trial
* Known or suspected allergy to insulin glargine or detemir
* Using other insulins, such as, bolus insulin or premixed insulin
* Sight or hearing impaired
* Pregnancy oor nursing of the intention of becoming pregnant or not using adequate contraceptive measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2006-10; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
In the time period 2400 to 0600 hours (the Basal Period) when post-meal food is least likely to affect the glucose level, detect the mean percentage pf time the glucose level is between 70-119 mg/dL

SECONDARY OUTCOMES:
Establish the mean percentage of time spent in the glucose ranges of 40-70 mg/dL, 120-179 mg/dL, 180-240 mg/dL and >240 mg/dL in the Basal Period and for the entire day, and the average glucose for the entire 24 hour period.

CONTACTS AND LOCATIONS:
Overall Officials: Allen B. King, MD, Principal Investigator — Diabetes Care Center
Locations (1):
- Diabetes Care Center, Salinas, California, United States

REFERENCES:
- [Background] Russell-Jones, D. et al. Diabetologia 2002;45(Suppl. 2):A51
- [Background] Boland E, Monsod T, Delucia M, Brandt CA, Fernando S, Tamborlane WV. Limitations of conventional methods of self-monitoring of blood glucose: lessons learned from 3 days of continuous glucose sensing in pediatric patients with type 1 diabetes. Diabetes Care. 2001 Nov;24(11):1858-62. doi: 10.2337/diacare.24.11.1858. PMID 11679447
- [Background] Bode BW, Gross TM, Thornton KR, Mastrototaro JJ. Continuous glucose monitoring used to adjust diabetes therapy improves glycosylated hemoglobin: a pilot study. Diabetes Res Clin Pract. 1999 Dec;46(3):183-90. doi: 10.1016/s0168-8227(99)00113-8. PMID 10624783
- [Background] Mastrototaro J. The MiniMed Continuous Glucose Monitoring System (CGMS). J Pediatr Endocrinol Metab. 1999;12 Suppl 3:751-8. No abstract available. PMID 10626266
- [Background] Metzger M, Leibowitz G, Wainstein J, Glaser B, Raz I. Reproducibility of glucose measurements using the glucose sensor. Diabetes Care. 2002 Jul;25(7):1185-91. doi: 10.2337/diacare.25.7.1185. PMID 12087017
- [Background] Gross TM, Mastrototaro JJ. Efficacy and reliability of the continuous glucose monitoring system. Diabetes Technol Ther. 2000;2 Suppl 1:S19-26. doi: 10.1089/15209150050214087. No abstract available. PMID 11469628
- [Background] Gross TM, Bode BW, Einhorn D, Kayne DM, Reed JH, White NH, Mastrototaro JJ. Performance evaluation of the MiniMed continuous glucose monitoring system during patient home use. Diabetes Technol Ther. 2000 Spring;2(1):49-56. doi: 10.1089/152091500316737. PMID 11467320
- [Background] King AB, Armstrong D. A comparison of basal insulin delivery: continuous subcutaneous insulin infusion versus glargine. Diabetes Care. 2003 Apr;26(4):1322. doi: 10.2337/diacare.26.4.1322. No abstract available. PMID 12663626
- [Background] King, AB, Armstrong, DU. Presentation at Diabetes Technology & Therapeutics Meeting, 2003, San Francisco
- [Background] Heise, T et al. Diabetes 2003;52(Suppl.1):A121